CLINICAL TRIAL: NCT00546039
Title: Effects of Synthetic Genistein Supplementation on Blood and Tissue Biomarkers in Patients With Localized Prostate Cancer
Brief Title: Synthetic Genistein (BONISTEIN™) in Patients Who Are Undergoing Surgery for Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Aker (Other)
Responsible Party: Bato Lazarevic MD, Aker University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: P2BV10
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate cancer; Localized prostatectomy; Laparoscopic prostatectomy; Chemoprevention; Genistein; BONISTEIN™
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Genistein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Genistein
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Genistein — Capsule, 30 mg, oral daily for 3 to 6 weeks
  Other Names: BONISTEIN™
  Arms: 1
Drug: Placebo — Capsule
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate safety and mechanisms of possible chemopreventive effects of synthetic genistein (BONISTEIN™) in patients with localized prostate cancer undergoing laparoscopic radical prostatectomy.

DETAILED DESCRIPTION:
In Norway prostate cancer is the most frequently diagnosed cancer in the male and represents the second most common cause of cancer death among men. Epidemiological studies have shown an association between decreased prostate cancer risk and increased soy consumption. Genistein is the dominating plasma and tissue isoflavone in soybean products, and it has been attributed several anti-cancer effects. BONISTEIN™ is a novel product, consisting of >99,5 % synthetic Genistein aglycone. Chemoprevention is the ability of certain molecules to inhibit (partially or totally) induction or progression of the disease. Our study population consists of men diagnosed with localized prostate cancer who have agreed to undergo radical prostatectomy. This provides adequate amount of benign, premalignant and malignant tissue for studying the effects of potential chemopreventive agents on biomarkers of cell growth and differentiation in the prostatic tissues with immunohistochemistry. Prostatic tissue cells will also be selected with Lacer Capture Microdissection (LCM) before analysis with semi-quantitative RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven prostate cancer clinical stage T1c or T2.
* Are to be treated by radical prostatectomy 3 to 6 weeks after consent.
* Have signed the informed consent form.

Exclusion Criteria:

* Have been on previous or concurrent hormonal therapy or chemotherapy.
* History of previous or other hormone dependent malignancies.
* Concomitant thyroid disease or are currently taking thyroid hormone replacement medication.
* On current high dose soy, micronutrient or herbal supplements.
* On soy or vegetarian nutrition or have any other extreme dietary habits.
* On oral anticoagulants.
* History of liver or pancreas diseases.
* History of hypersensitivity to Genistein or soy containing products.
* Have a malabsorption condition which might interfere with absorption of the investigational product.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Modulation of biomarkers: PSA, Testosterone, STAMP1, STAMP2, NKX3A and KLK4, p21, p27, p53, bcl-2, bax, Ki67, CgA and NSE in blood and/or prostate tissue. | 3 to 6 weeks

SECONDARY OUTCOMES:
Modulation of prostate cancer grade, volume and Gleason score. Safety parameters (blood, electrolytes, liver, pancreas, lipids, thyroid and sexual hormones). Plasma and tissue concentrations of BONISTEIN™. | 3 to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steinar J Karlsen, MD, PhD, Study Director — Aker University Hospital, Oslo Urological Universityclinic; Bato Lazarevic, MD, Principal Investigator — Aker University Hospital, Oslo Urological Universityclinic
Locations (1):
- Aker University Hospital, Oslo, Norway

REFERENCES:
- See also: Homepage Aker University Hospital — http://www.aus.no/